CLINICAL TRIAL: NCT04325308
Title: Early Life Protein-enriched Human Milk Diets to Increase Lean Body Mass Accretion and Diversity of the Gut Microbiome in Extremely Preterm Infants: a Randomized Trial
Brief Title: Early Protein Supplementation in Extremely Preterm Infants Fed Human Milk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ariel A. Salas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 300005089; K23HD102554 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Prematurity; Extreme; Feeding Disorder Neonatal; Breast Milk Expression; Growth Failure; Microbial Colonization
MeSH Terms: conditions — Premature Birth; Breast Milk Expression; Failure to Thrive; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Caregivers and primary outcome evaluators will be masked. Nutrition room staff not involved in patient care will be responsible for determining participant allocation to one of the supplementation groups by opening sequentially numbered sealed envelopes, dispensing feeding syringes with the allocated human milk diet (protein-enriched or usual), and masking caregivers administering the assigned dietary intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-enriched human milk diet (Experimental): Infants in this group will receive protein-enriched expressed human milk or donor human milk during the first 2 weeks after birth.
  Interventions: Procedure: Protein-enriched human milk diet
- Usual human milk diet (Active Comparator): Infants in this group will receive either expressed human milk or donor human milk during the first 2 weeks after birth.
  Interventions: Procedure: Usual human milk diet

INTERVENTIONS:
Procedure: Protein-enriched human milk diet — 1.2 g of human-based protein will be added to each 100 ml of human milk administered
  Arms: Protein-enriched human milk diet
Procedure: Usual human milk diet — Human-based protein will not be added to the human milk administered.
  Arms: Usual human milk diet

SUMMARY:
The central hypothesis of this clinical trial is that, in extremely preterm infants, protein-enriched human milk diets compared to usual human milk diets during the first 2 weeks after birth increase fat-free mass (FFM)-for-age Z scores and promote maturation of the gut microbiome at term corrected age.

DETAILED DESCRIPTION:
Masked randomized clinical trial in which extremely preterm infants fed human milk will be randomly assigned to receive either a protein-enriched diet (intervention group) or a usual diet (control group) within the first 96 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 28 weeks of gestation
* Postnatal age < 96 hours

Exclusion Criteria:

* Congenital malformations
* Chromosomal anomalies
* Terminal illness needing to limit or withhold support

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tucker MJ, Jeffcoat SH, Argent T, Travers CP, Salas AA. Severity of Bronchopulmonary Dysplasia in Infants Born Extremely Preterm and Randomized to Early Human Milk Fortification with a Donor Milk-Derived Fortifier for 2 Weeks. J Pediatr. 2025 Dec;287:114750. doi: 10.1016/j.jpeds.2025.114750. Epub 2025 Jul 24. PMID 40714049
- [Result] Salas AA, Gunawan E, Nguyen K, Reeves A, Argent V, Finck A, Carlo WA. Early Human Milk Fortification in Infants Born Extremely Preterm: A Randomized Trial. Pediatrics. 2023 Sep 1;152(3):e2023061603. doi: 10.1542/peds.2023-061603. PMID 37551512

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Started | 75 | 75
Completed | 52 | 53
Not Completed | 23 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Median (Inter-Quartile Range); unit: weeks of gestation] | 26 [24 to 27] | 26 [24 to 27] | 26 [24 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 29 | 72
  Male | 32 | 46 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 70 | 68 | 138
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 38 | 83
  White | 29 | 36 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Fat-free Mass(FFM)-For-age Z-score
Description: Estimated by air displacement plethysmography. FFM measurements were converted into Z-scores using updated, sex-specific reference curves of body composition in preterm infants (Norris et al, 2019). A Z-score of 0 represents the population mean. Z-score values closer to 0 represent a better outcome. No relevant thresholds have been defined.
Time Frame: 36 weeks or hospital discharge, up to 120 days following birth, whichever is longer
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 52 | 53
Z-score | -1.7 (1.4) | -1.6 (1.5)

2. Secondary Outcome: Fat Mass(FM)-For-age Z-score
Description: Estimated by air displacement plethysmography. FM measurements were converted into Z-scores using updated, sex-specific reference curves of body composition in preterm infants (Norris et al, 2019). A Z-score of 0 represents the population mean. Z-score values closer to 0 represent a better outcome. No relevant thresholds have been defined.
Time Frame: 36 weeks or hospital discharge, up to 120 days following birth, whichever is longer
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 52 | 53
Z-score | 1.0 (1.1) | 1.3 (1.2)

3. Secondary Outcome: Body Fat(BF)-For-age Z-score
Description: Body fat estimated by air displacement plethysmography. BF measurements were converted into Z-scores using updated, sex-specific reference curves of body composition in preterm infants (Norris et al, 2019). A Z-score of 0 represents the population mean. Z-score values closer to 0 represent a better outcome. No relevant thresholds have been defined.
Time Frame: 36 weeks or hospital discharge, up to 120 days following birth, whichever is longer
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 52 | 53
Z-score | 1.8 (1) | 1.9 (1.2)

4. Secondary Outcome: Anthropometric Measurements
Description: Weight, length, and head circumference measurements. Measurements were converted into Z-scores based on Fenton growth curves (2013). They were calculated at birth and at 36 weeks. This outcome represents the change in weight, length, and head circumference Z-score during the course of the study (i.e., the Z-score at birth was subtracted from the Z-score at 36 weeks).
  A value of 0 represents that the infant's Z-score is the same at the beginning and the end of the study. Positive values indicate the increase in the infant's Z-score during the study; negative values indicate the decrease in the infant's Z-score during the study.
Time Frame: Birth to 36 weeks postmenstrual age or hospital discharge (whichever occurred first)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 65 | 63
Z-score
  Weight | -1.0 (0.7) | -1.2 (0.8)
  Length | -1.5 (1.0) | -1.9 (1.3)
  Head circumference | -0.9 (0.8) | -1.3 (1.1)

5. Secondary Outcome: Growth Rate
Description: Weight gain in g/kg/day
Time Frame: Birth to 36 weeks postmenstrual age or hospital discharge (whichever occurred first)
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 65 | 63
g/kg/day | 14.7 (2.5) | 13.9 (2.5)

6. Secondary Outcome: Number of Participants With Postnatal Growth Failure
Description: Diagnosis of growth failure (weight < 10th percentile using the 2013 Fenton growth curves)
Time Frame: 36 weeks or hospital discharge (whichever occurred first)
Measure: Count of Participants; unit: Participants
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 65 | 63
Participants | 31 | 30

7. Secondary Outcome: Number of Participants With Diagnosis of Necrotizing Enterocolitis
Description: Diagnosis of necrotizing enterocolitis stage 2 or 3
Time Frame: From birth up to 120 days following birth
Measure: Count of Participants; unit: Participants
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 75 | 75
Participants | 1 | 3

8. Secondary Outcome: Number of Participants With Diagnosis of Intestinal Perforation
Description: Diagnosis of intestinal perforation
Time Frame: From birth up to 120 days following birth
Measure: Count of Participants; unit: Participants
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 75 | 75
Participants | 5 | 4

9. Secondary Outcome: Death
Description: Death prior to 121 days of life
Time Frame: Birth to 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 65 | 63
Participants | 6 | 5

10. Secondary Outcome: Culture-proven Sepsis
Description: Diagnosis of sepsis with positive blood cultures
Time Frame: Birth to 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 75 | 75
Participants | 22 | 16

11. Secondary Outcome: Number of Days Alive and Receiving Full Enteral Feeding
Description: Time to full enteral feeding days
Time Frame: Birth to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 68 | 71
days | 18 [11 to 21] | 14 [5 to 18]

12. Secondary Outcome: Number of Episodes of Feeding Intolerance
Description: Interruption or cessation of enteral feeds for a period greater than 12 hours for abnormal abdominal examination
Time Frame: Birth to 28 days
Population: Not collected
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Duration of Hospital Stay in Days
Description: From day of admission to day of hospital discharge to home
Time Frame: Birth to 120 days or discharge, whichever occurs first
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 69 | 70
days | 107 [87 to 120] | 107 [79 to 120]

14. Secondary Outcome: Serum BUN
Description: Highest serum BUN value in the first 28 days after birth
Time Frame: Birth to 28 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
Number analyzed (Participants) | 69 | 69
mg/dL | 33 (24) | 37 (31)

15. Other Pre Specified Outcome: Changes in Intestinal Microbiome
Description: Determined by molecular analyses of fecal samples
Time Frame: Birth to 36 weeks postmenstrual age
Reporting Status: Not Posted, anticipated posting 2026-05

16. Other Pre Specified Outcome: Cognitive Outcomes
Description: Determined by Bayley assessment
Time Frame: 2 years of corrected age
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: From birth up to 120 days following birth
Arm/Group | Protein-enriched Human Milk Diet | Usual Human Milk Diet
All-Cause Mortality (participants affected / at risk) | 6/75 | 5/75
Serious Adverse Events (participants affected / at risk) | 6/75 | 4/75
Other Adverse Events (participants affected / at risk) | 31/75 | 30/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Protein-enriched Human Milk Diet (N=75) | Usual Human Milk Diet (N=75)
Necrotizing enterocolitis (Gastrointestinal disorders) | 1 | 3
Spontaneous intestinal perforation (Gastrointestinal disorders) | 5 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Protein-enriched Human Milk Diet (N=75) | Usual Human Milk Diet (N=75)
Growth failure (General disorders) | 31 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04325308/Prot_SAP_000.pdf